CLINICAL TRIAL: NCT00526344
Title: Bronchoscopy and Bronchial Biopsies. Sub-study of: Characteristics of Asthma Remissions
Brief Title: Bronchoscopy With Bronchial Biopsies Sub-study of: Persistence of Airway Inflammation and Remodeling in Asthma Remission
Status: Withdrawn | Type: Observational
Why Stopped: No funding, study not done
Sponsor: Laval University (Other)
Responsible Party: Louis-Philippe Boulet, Laval Hospital
Other Study IDs: HL-07- sep-biop
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Asthma
Keywords: remission of asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue (bronchial biopsies)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Subjects with complete remission of asthma
- 2: Subjects with symptomatic remission of asthma
- 3: Subjects with asthma
- 4: Healthy controls

SUMMARY:
This study aims at determining the patterns of asthma remission, the prevalence of these different patterns and the various factors associated with such remissions and possible recurrences of asthma, in order to determine the mechanisms involved in these processes.

We therefore want to document these specificities in studying biopsies of subjects in complete remission of their asthma and those in only symptomatic remission of their asthma, in comparison with mildly symptomatic asthmatic subjects and healthy controls.

DETAILED DESCRIPTION:
Primary Outcome Measures :

Airway inflammation and remodeling: in bronchial biopsies

Secondary Outcome Measures:

Comparisons of bronchial biopsy features between groups:

* Bronchial epithelial morphology
* Bronchial mucosa (smooth muscle, reticular basement membrane, submucosal gland,...)

ELIGIBILITY:
Inclusion Criteria:

* In remission of their asthma: absence of respiratory symptoms, no rescue asthma medication need and (for complete remission) an optimal pulmonary function (FEV1 > 90%) and normal PC20 methacholine for more than two years (with no current treatment).
* With a proven past history of asthma from medical files (reversible airway obstruction (> 12% FEV1 after bronchodilator or 20% by other means) proven by spirometry, PEF measures or methacholine challenge according to current criteria + previous symptoms and asthma medication use), having no more asthma symptoms and not having used asthma medication for more than 2 years.
* Agree to sign the consent form.
* No other condition that could interfere with the study measurements.

Exclusion Criteria:

* Subjects using inhaled or oral anti-inflammatory agents.
* FEV1 < 1.2 L.
* Unable to adhere to the protocol requirements.
* Other current respiratory disease
* Upper or lower respiratory tract infection or use of antibiotics < 1 month.
* Use of oral corticosteroids within the last 3 months.
* Signs or symptoms of progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with current asthma or in remission of asthma from primary care clinics will be allowed to participate to this study. Healthy subjects will also be invited by advertisements in newspapers to volunteer for this study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2007-09; Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulat, MD, Principal Investigator — Hôpital Laval
Locations (1):
- Centre de Recherche, Hôpital Laval, Québec, Quebec, Canada